CLINICAL TRIAL: NCT01717898
Title: A Multicenter Phase I/II Trial of Abiraterone Acetate + BEZ235 in Metastatic, Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Dose limiting toxicities on lowest dose level
Sponsor: Charles Ryan (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Charles Ryan, Associate Professor of Clinical Medicine & Urology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF CC#125510
Record Dates: First submitted 2012-10-23; First posted 2012-10-31 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Castrate-resistant Prostate Cancer
Keywords: Castrate-resistant prostate cancer
MeSH Terms: interventions — dactolisib; Prednisone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone/prednisone + BEZ235 (Experimental): In Phase I, a dose escalation of BEZ235 will be performed using a standard 3 + 3 design to determine the maximum tolerated dose (MTD) of BEZ235 given in combination with continuous fixed doses of Abiraterone Acetate and prednisone. This BEZ235 dose will be used in the phase II portion of the study.
  Interventions: Drug: BEZ235; Drug: Prednisone; Drug: Abiraterone acetate

INTERVENTIONS:
Drug: BEZ235 — BEZ235 - 200 mg, 300 mg, or 400 mg; po, BID. BEZ235 will be supplied in 200 mg, 300 mg, and 400 mg sachets packaged in boxes.
Drug: Prednisone — 10/mg po daily. Prednisone can be modified at the investigator's discretion, but should not be discontinued.
Drug: Abiraterone acetate — 1000 mg, po. Abiraterone Acetate is supplied in 250 mg white tablets, four tablets are to be taken with a full glass of water on an empty stomach once daily.
  Other Names: CB7630

SUMMARY:
There will be two parts to this clinical research study. The purpose of each part is:

* Phase 1: This part of the study will determine what dose of BEZ235 is safe to give with a standard dose of abiraterone acetate and prednisone by administering different doses of BEZ235. This will help to find out what effects, good and/or bad, this combination has on CRPC.
* Phase 2: This part of the study will measure the treatment effect of the combination of BEZ235 and abiraterone acetate/prednisone on CRPC.

DETAILED DESCRIPTION:
Prostate Cancer Overview:

Prostate cancer is the second most common cancer in men representing approximately 30% of all cancers diagnosed in men. When confined to the prostate gland the disease is curable with local therapy. However approximately 50% of men fail local therapy and develop incurable metastatic disease. Androgen deprivation (AD) therapy remains the mainstay of treatment, not only for advanced disease but also in the adjuvant and neo-adjuvant settings. Androgen deprivation therapy induces a remission in 80 to 90% of patients with advanced disease and results in a median progression-free survival of 12 to 33 months, at which time an androgen-independent phenotype usually emerges. This accounts for the median overall survival of 23 to 37 months from the initiation of androgen deprivation.

Androgen deprivation can be achieved surgically with orchiectomy, or using some form of drug treatment. Current approaches to AD utilize leutinizing hormone releasing hormone (LHRH) agonists. These act by continuous stimulation of the anterior pituitary resulting in inhibition of leutinizing hormone (LH) secretion, and hence a fall in testicular production of testosterone. Although AD is clinically effective in the majority of patients, studies have shown that extratesticular sources of testosterone represent an important alternative source of androgen stimulation in a significant proportion of prostate cancer patients. As much as 10% of baseline circulating testosterone remains in castrate men, due to the peripheral conversion of adrenal steroids to testosterone. Increased levels of androgen receptor confer resistance to antiandrogens in prostate cancer xenograft models. This could result in amplified signal output from circulating low levels of adrenal androgens and suggests a role for agents that target the adrenal androgen synthesis pathway.

As prostate cancer progresses to castration-resistant prostate cancer genetic events accumulate. One of the most consistent genetic findings in CRPC is amplification and over-expression of the androgen receptor (AR). Multiple groups have demonstrated that up-regulation of AR expression along with de novo synthesis of androgens by the adrenals and/or prostate cancer cells themselves is perhaps the most common mechanism by which prostate cancer cells progress despite castrate levels of circulating testosterone. This underlying biology is likely the mechanism explaining the recent success of Abiraterone Acetate.

An important genetic event found to be associated with progression of prostate cancer is loss of heterozygosity and subsequent homozygous deletion at the 10q23 locus containing the PTEN tumor suppressor gene. PTEN functions, in part, as a negative regulator of the phosphatidylinositol 3' (PI3) kinase - AKT pathway. Targeting the PI3K pathway and/or downstream targets of PI3K has been recognized as an important therapeutic strategy for some time. An important aspect of PI3K signaling is the PTEN mutation and the downstream events associated with PI3K signaling are not mutually exclusive with the aforementioned AR signaling pathway aberrancies that have yielded important therapeutic consequences. Preclinical data has demonstrated that PI3K inhibition upregulates AR expression, but that the net effect is antiproliferative and that concomitant anti androgen therapy is synergistic.

Introduction to BEZ235 and Abiraterone Acetate:

Preclinical data has demonstrated that PI3K inhibition upregulates AR expression, and that concomitant anti-androgen therapy has synergistic anti-tumor effects with PI3K inhibition. This study seeks to enhance the efficacy of Abiraterone Acetate in CRPC by concomitantly targeting PI-3Kinase activity with the novel agent BEZ-235.

BEZ235 is a potent pan-class I PI3K and mammalian target of rapamycin (mTOR) inhibitor belonging to the class of imidazoquinoline derivatives. BEZ235 is the investigational agent utilized in this study.

Abiraterone Acetate is now considered a standard of care for the treatment of Castration Resistant Prostate Cancer (CRPC) following docetaxel, and is likely to be considered such in the pre-chemotherapy setting based on recent results. Despite benefits in survival resistance to this therapy develops in virtually all patients.

Study rationale and purpose:

It is hypothesized that signaling through the PI3Kinase pathway is a major mechanism of resistance to Abiraterone Acetate therapy (and castration based therapy in general) and that inhibition of this pathway will enhance the clinical benefit of Abiraterone Acetate.

The addition of BEZ 235 to Abiraterone Acetate provides an opportunity to test if inhibition of PI3K along with TORC1 will attenuate the survival mechanisms co-opted by CRPC when treated with Abiraterone Acetate. We will conduct a Phase I study to determine the MTD for this combination and use that dose for this Phase II study. Biopsies of metastatic disease prior to and during treatment with BEZ235 plus Abiraterone Acetate will allow for the determination if mutations in the PTEN and/or PI3kinase axis in biopsied tumors are associated with response to therapy with the combination of BEZ235 and Abiraterone Acetate.

While PSA decline remains an imperfect surrogate marker for overall survival it remains a useful means of determining whether a positive clinical "signal" exists for a given treatment strategy and can be an efficient means of determining if an approach could proceed to more definitive testing according the standards of the Prostate Cancer Working Group 2 (PCWG2).

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. Patient has provided a signed study Informed Consent Form prior to any screening procedure.
2. Patient is ≥ 18 years of age on the day of consenting to the study.
3. Patients must have histologically confirmed adenocarcinoma of the prostate.
4. Radiographic evidence of disease (bone scan, CT scan, ultrasound or MRI acceptable) that is amenable to image-guided biopsy must be present.
5. Patients must have castrate levels of testosterone (< 50 ng/dL) on GnRH analogues or have had prior orchiectomy. GnRH analogues must be continued while on study.
6. Progressive disease as demonstrated by a rising PSA or radiographic progression per PCWG2 criteria.
7. Asymptomatic or minimally symptomatic disease: No use of opiate analgesics (EXCLUDING codeine or dextromethorphan) for cancer related pain within 28 days of day 1, cycle 1.
8. Phase II Cohort 1: No prior Abiraterone Acetate therapy
9. Phase II Cohort 2: Immediate prior Abiraterone Acetate therapy is required. No intervening therapy is allowed between Abiraterone Acetate therapy and study therapy.
10. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
11. Men of reproductive potential who have not had a radical prostatectomy must agree to use an effective contraceptive method. Patients who have had a prostatectomy are sterile and do not need to use contraception.
12. Patient has adequate bone marrow and organ function as shown by:

    * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
    * Platelets ≥ 100 x 109/L
    * Hemoglobin (Hgb) ≥ 9.0 g/dL
    * INR ≤ 2
    * Serum creatinine ≤ 1.5 x ULN
    * Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
    * AST and ALT ≤ 3 x ULN (or ≤ 5.0 x ULN if hepatic metastases are present)
    * Fasting plasma glucose (FPG) ≤ 140mg/dL [7.8 mmol/L]
    * HgbA1c ≤8% (Patients with diabetes mellitus not actively being treated and patients with an HgbA1c level between 7-8% will be required to have home glucose monitoring three times weekly during the first cycle. Patients may also be referred to a diabetes specialist as indicated.)

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Patient has received previous treatment with PI3K and/or mTOR inhibitors.
2. Phase II Cohort 1: Prior Abiraterone Acetate therapy is an exclusion
3. Prior therapy with any of the following for >1 month: MDV-3100, Orteronel, ketoconazole or other drugs given with the intention to inhibit CYP 17.
4. Patient has active uncontrolled or symptomatic CNS metastases. Note: A patient with controlled and asymptomatic CNS metastases may participate in this trial. As such, the patient must have completed any prior treatment for CNS metastases > 90 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
5. Patient has a concurrent malignancy or has had a malignancy in the last 3 years prior to start of study treatment (with the exception of adequately treated basal or squamous cell carcinoma or cervical carcinoma in situ).
6. Patient has received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug or has not recovered from side effects of such therapy.
7. Patient has had major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery.
8. Patient has active cardiac disease including any of the following:

   * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * QTcF > 480 msec on screening ECG
   * Unstable angina pectoris
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with documented compromise in cardiac function
   * Symptomatic pericarditis
9. Patient has a history of cardiac dysfunction including any of the following:

   * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function.
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
10. Family history of congenital long or short QT, or known history of QT/QTc prolongation or Torsades de Pointes (TdP).
11. Patient with medically documented history of active major depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation.
12. Active or uncontrolled infection of hepatitis B or hepatitis C.
13. Inadequately controlled hypertension (i.e., SBP > 180 mmHg or DBP > 100 mmHg).
14. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235 (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea grade ≥ 2, malabsorption syndrome or small bowel resection).
15. Use of any chemotherapy, investigational agents, immunotherapy, or hormonal therapy other LHRH agonists within 28 days of the start of treatment on protocol. Use of bone targeted agents including bisphosphanates and RANK ligand inhibitors is allowed if on stable dose; Xgeva or Zometa cannot be started within 28 days of initiating study therapy.
16. Systemic corticosteroids except as part of on label treatment prostate cancer regimens.

    Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed.
17. Patient is undergoing active treatment for diabetes mellitus.
18. Patient is being treated at start of study treatment with any of the following drugs:

    * Drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications (see Appendix 1 for a list of prohibited CYP3A4 inhibitors and inducers)
    * Drugs with a known risk to induce Torsades de Pointes (see Appendix 3 for a list of prohibited drugs)
    * Warfarin and coumadin analogues
19. Patient is consuming Seville oranges, grapefruit, grapefruit hybrids, pomelos and exotic citrus fruits (as well as their juices) during the last 7 days prior to start of treatment. Regular orange juice is permitted.
20. Immunocompromised patients, including known seropositivity for HIV (testing is not mandatory).
21. Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate his participation in the clinical study (e.g. uncontrolled diabetes, chronic pancreatitis, active chronic hepatitis etc.).
22. Patient is not able to understand or to comply with study instructions and requirements or has a history of non-compliance to medical regimen.
23. Patients in whom, in the opinion of the treating physician, should receive cytotoxic chemotherapy with docetaxel.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2013-09-03 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Wei XX, Hsieh AC, Kim W, Friedlander T, Lin AM, Louttit M, Ryan CJ. A Phase I Study of Abiraterone Acetate Combined with BEZ235, a Dual PI3K/mTOR Inhibitor, in Metastatic Castration Resistant Prostate Cancer. Oncologist. 2017 May;22(5):503-e43. doi: 10.1634/theoncologist.2016-0432. Epub 2017 Mar 17. PMID 28314838

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: BEZ235 200 mg: Dose level 1:
  200 mg BEZ235 orally (PO) twice a day (BID)
  Prednisone: 10/mg PO daily
  Abiraterone acetate: 1000 mg, PO daily
- Phase I: BEZ235 300 mg: Dose level 2:
  300 mg BEZ235 orally (PO) twice a day (BID)
  Prednisone: 10/mg PO daily.
  Abiraterone acetate: 1000 mg, PO daily
- Phase I: BEZ235 400 mg: Dose level 3:
  400 mg BEZ235 orally (PO) twice a day (BID)
  Prednisone: 10/mg po daily. Prednisone can be modified at the investigator's discretion, but should not be discontinued.
  Abiraterone acetate: 1000 mg, po.
- Phase II: Phase II:
  BEZ235 at MTD
  Prednisone 5 mg twice daily
  Abiraterone 1,000 mg daily
Period: Overall Study
Arm/Group | Phase I: BEZ235 200 mg | Phase I: BEZ235 300 mg | Phase I: BEZ235 400 mg | Phase II
Started | 6 | 0 (Study was terminated during Phase I, Dose level 1 due to toxicity.) | 0 (Study was terminated during Phase I, Dose level 1 due to toxicity.) | 0 (Study was terminated during Phase I, Dose level 1 due to toxicity.)
Completed | 0 (Study was terminated during Phase I, Dose level 1 due to toxicity.) | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone/Prednisone + BEZ235
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 71 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Dose Limiting Toxicities When Combining BEZ235 With Abiraterone Acetate (Phase I).
Time Frame: Beginning of study up to 15 months
Population: Study was terminated during Phase I, Dose level 1 due to toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: BEZ235 200 mg: Dose level 1:
  200 mg BEZ235 orally (PO) twice a day (BID)
  Prednisone: 10/mg PO daily Prednisone can be modified at the investigator's discretion, but should not be discontinued.
  Abiraterone acetate: 1000 mg, PO daily
- Phase I: BEZ235 300 mg: Dose level 2:
  300 mg BEZ235 orally (PO) twice a day (BID)
  Prednisone: 10/mg PO daily. Prednisone can be modified at the investigator's discretion, but should not be discontinued.
  Abiraterone acetate: 1000 mg, PO daily
Arm/Group | Phase I: BEZ235 200 mg | Phase I: BEZ235 300 mg | Phase I: BEZ235 400 mg | Phase II
Number analyzed (Participants) | 6 | 0 | 0 | 0
Participants | 3 | 0 | 0 | 0

2. Primary Outcome: Anti-tumor Responses as Defined by a Decline in PSA of > 50%
Description: Anti-tumor responses as defined by a decline in PSA of > 50% following 12 weeks of therapy to the combination of Abiraterone Acetate plus BEZ-235 occur in a cohort of patients who have received prior therapy with Abiraterone Acetate therapy
Time Frame: From day 1 of therapy initiation up to 12 weeks
Population: Study was terminated during Phase I, Dose level 1 due to toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BEZ235 200 mg | Phase I: BEZ235 300 mg | Phase I: BEZ235 400 mg | Phase II
Number analyzed (Participants) | 6 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Response Proportion as Defined by a Decline in PSA of > 50%
Description: Response proportion as defined by a decline in PSA of > 50% following 12 weeks of therapy for patients treated with the combination of BEZ235 and Abiraterone Acetate plus Prednisone (Phase II outcome measure).
  Study was terminated during Phase I, Dose level 1 due to toxicity, therefore no Phase II data is available.
Time Frame: From day 1 of therapy initiation up to 12 weeks
Population: Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase I: BEZ235 200 mg | Phase I: BEZ235 300 mg | Phase I: BEZ235 400 mg | Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Maximum Tolerated Dose for BEZ235 + Abiraterone Acetate (Phase I).
Description: Maximum Tolerated Dose (MTD) for BEZ235 + Abiraterone Acetate (to be determined during Phase I). The MTD of BEZ235 will be the dose when given in combination results in less than 33% dose limiting toxicities (DLT).
Time Frame: Beginning of study up to 15 months
Population: Dose could not be determined. Study was terminated during Phase I, Dose level 1 due to toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: BEZ235 200 mg | Phase I: BEZ235 300 mg | Phase I: BEZ235 400 mg | Phase II
Number analyzed (Participants) | 6 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Trough Concentrations of BEZ235 and Abiraterone Acetate Plus Prednisone When Used in Combination
Description: Trough concentrations of BEZ235 and Abiraterone Acetate plus Prednisone when used in combination during Phase I.
Time Frame: Beginning of study up to 15 months
Population: Concentrations could not be determined. Study was terminated during Phase I, Dose level 1 due to toxicity.
Groups:
- BEZ235: Trough concentration of BEZ235 when used in combination with Abiraterone plus Prednisone.
- Abiraterone Acetate: Trough concentration of Abiraterone acetate when used in combination with BEZ235 plus Prednisone.
Arm/Group | BEZ235 | Abiraterone Acetate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS) in Phase II
Description: Progression Free Survival (PFS) of the combination of BEZ235 plus Abiraterone Acetate/prednisone as determined by Prostate-Specific Antigen Working Group 2 criteria (PSAWG2 ) during Phase II.
Time Frame: Beginning of Phase II up to 15 months
Population: PFS in Phase II could not be determined. Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase II
Number analyzed (Participants) | 0

7. Secondary Outcome: Determination of the Time to PSA Progression in Phase II
Description: Determination of the time to PSA progression in Phase II based on PSAWG2 criteria.
Time Frame: Beginning of Phase II up to 15 months
Population: Time to PSA progression could not be determined. Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase II
Number analyzed (Participants) | 0

8. Secondary Outcome: Objective Response Rate (ORR) in Phase II
Description: Proportion of patients achieving an objective response to BEZ235 + Abiraterone Acetate/prednisone according to RECIST criteria.
Time Frame: From beginning of Phase II up to 15 months
Population: ORR could not be determined. Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase II
Number analyzed (Participants) | 0

9. Secondary Outcome: Safety of BEZ235 and Abiraterone Acetate Plus Prednisone When Used in Combination
Description: Number of reported Adverse Events in BEZ235 and Abiraterone Acetate plus Prednisone when used in combination (Phase II).
Time Frame: Beginning of Phase II up to 15 months
Population: No Adverse Events were collected in Phase II. Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase II
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Determination of Whether the Pre-treatment Status of pS6, pAKT, p4EBP1 and PTEN, Determined by IHC in the Optional Biopsies of Metastatic Tumors, Are Associated With Response to BEZ235 Plus Abiraterone Acetate/Prednisone.
Time Frame: post study
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Determination of Whether Specific Pathway Changes Are Predictive of Clinical Benefit (Improved PFS) or Resistance Prior to Treatment or During Treatment Using Microarray Analysis.
Time Frame: post study
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Phase I: Abiraterone/Prednisone + BEZ235 200 mg: Study was terminated during Phase I, Dose level 1 due to toxicity.
Arm/Group | Phase I: Abiraterone/Prednisone + BEZ235 200 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Abiraterone/Prednisone + BEZ235 200 mg (N=6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Abiraterone/Prednisone + BEZ235 200 mg (N=6)
Anemia (Blood and lymphatic system disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Malaise (General disorders) | 1
Creatinine increased (Endocrine disorders) | 1
Serum amylase increased (Endocrine disorders) | 1
Weight loss (General disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
Study got terminated due to safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No